CLINICAL TRIAL: NCT02501343
Title: Alkaline Diet for Insulin Sensitivity
Acronym: ADIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Dorit Samocha-Bonet, Leader, Clinical Insulin Resistance Group, Diabetes and Metabolism Division, Garvan Institute of Medical Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ADIS (SVH 14/157)
Record Dates: First submitted 2015-07-13; First posted 2015-07-17 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Dysglycemia; Type 2 Diabetes Mellitus
Keywords: Glucose metabolism; Potential renal acid load; Postprandial glycemia; Body acid-base homeostasis; Sodium bicarbonate
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium bicarbonate (Experimental): High acid load meal (Western style meal) with Sodium bicarbonate (Sodibic 840mg*2)
  Interventions: Drug: Sodium Bicarbonate Oral Capsule
- Placebo (Placebo Comparator): High acid load meal (Western style meal) with sodibic-matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Bicarbonate Oral Capsule — Sodium bicarbonate 1680 mg will be administered prior to the meal
  Other Names: Sodibic capsules (Aspen Australia, NSW, Australia)
  Arms: Sodium bicarbonate
Drug: Placebo — Sodibic-matching placebo (Stenlake Compounding Chemist, NSW, Australia) will be administered prior to the meal on a different day 1 to 2 weeks apart
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the effect of increasing the body pH acutely with an alkaline medication (sodium bicarbonate, NaHCO3, sodibic) on glucose metabolism post meal in non diabetic subjects with normal renal function.

The investigators aim to determine whether there is an acute reduction in venous blood pH following a typical Western-style (high acid load) breakfast in healthy men and women, and whether this effect is attenuated by the concurrent administration of an alkaline medication. The effect on glucose metabolism, hunger/satiety and arterial stiffness post meal will be assessed.

DETAILED DESCRIPTION:
The aim of the study is to test the effect of increasing the body pH acutely with an alkali (NaHCO3) prior to a high acid load meal on glucose metabolism in non-diabetic men and women.

This is a double-blind placebo-controlled randomised study with a crossover design.

Study Procedures:

Two (2) meal studies will be performed 1 to 2 weeks apart. Studies will include collecting fasting blood to assess circulating glucose, insulin, C-peptide, free fatty acids, glucagon-like peptide-1, acid/base markers, including electrolytes (EUC) and venous blood pH. Participants will then be either administered sodibic (1680 mg) or matching placebo and a standardised Western style/high acid load meal. Investigators and participants will be blinded to the intervention. Blood will be drawn every 15 min in the first hour and then every 30 min for 3 hours in total. Arterial stiffness and appetite score will be evaluated at ½ h intervals.

Sample size: 30

sample size calculation: To detect a difference in area under the curve (AUC) of venous blood pH with a paired crossover design, 32 individuals will be required with statistical power 1-β>0.8 (allowing for drop-out).

statistical considerations: Differences between AUC of outcome measures post sodium bicarbonate vs. placebo will be tested using paired t-tests. Two-way repeated measure ANOVA tests will be conducted to assess differences in the response to the meal with sodium bicarbonate vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 22-65
* Disease status: Healthy.
* Laboratory parameters: Fasting plasma glucose <7 mmol/L, HbA1c <6.5% (48 mmol/mol).
* Willingness to give written informed consent and willingness to participate and comply with the study.

Exclusion Criteria:

* Individuals with a personal history of diabetes, hypertension, cardiovascular disease, kidney disease, respiratory disease or inflammatory disease.
* Individuals treated with medications known to affect insulin sensitivity.
* Individuals with fasting plasma glucose ≥7 mmol/L, HbA1c ≥6.5% (48 mmol/mol).
* Individuals with an unstable body weight in the past 3 months (+/- 2 kg or more).
* Individuals with a history of a psychological illness or condition that may interfere with the participant's ability to understand the requirements of the study.
* Individuals who smoke.
* Individuals who consume more than 40 g of alcohol daily.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in venous blood pH | Baseline (fasting) and 3 hours post meal
  The investigators aim is to determine whether venous blood pH decreases after a high acid load meal, and whether this effect is attenuated by administration of sodium bicarbonate prior to a mixed meal study

SECONDARY OUTCOMES:
Changes in glycemic response to the meal | Baseline (fasting) and 3 hours post meal
  Postprandial glucose excursion will be compared between sodium bicarbonate and placebo
Changes in insulin response to the meal | Baseline (fasting) and 3 hours post meal
  Postprandial insulin excursion will be compared between sodium bicarbonate and placebo
Changes in arterial stiffness | Baseline (fasting) and 3 hours post meal
  Postprandial arterial stiffness (measured by the augmentation index derived from Sphygmocore, Atcor Medical, Australia) will be compared between sodium bicarbonate and placebo
Changes in hunger and satiety scores | Baseline (fasting) and 3 hours post meal
  Postprandial hunger and satiety will be compared between sodium bicarbonate and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Samocha-Bonet, BSc(Hons) MSc(Hons) PhD, Principal Investigator — Garvan Institute of Medical Research
Locations (1):
- Garvan Institute of Medical Research, Darlinghurst, New South Wales, Australia

REFERENCES:
- [Background] DeFronzo RA, Beckles AD. Glucose intolerance following chronic metabolic acidosis in man. Am J Physiol. 1979 Apr;236(4):E328-34. doi: 10.1152/ajpendo.1979.236.4.E328. PMID 434194
- [Background] Fagherazzi G, Vilier A, Bonnet F, Lajous M, Balkau B, Boutron-Rualt MC, Clavel-Chapelon F. Dietary acid load and risk of type 2 diabetes: the E3N-EPIC cohort study. Diabetologia. 2014 Feb;57(2):313-20. doi: 10.1007/s00125-013-3100-0. PMID 24232975
- [Background] Reaich D, Graham KA, Channon SM, Hetherington C, Scrimgeour CM, Wilkinson R, Goodship TH. Insulin-mediated changes in PD and glucose uptake after correction of acidosis in humans with CRF. Am J Physiol. 1995 Jan;268(1 Pt 1):E121-6. doi: 10.1152/ajpendo.1995.268.1.E121. PMID 7840169
- [Background] Souto G, Donapetry C, Calvino J, Adeva MM. Metabolic acidosis-induced insulin resistance and cardiovascular risk. Metab Syndr Relat Disord. 2011 Aug;9(4):247-53. doi: 10.1089/met.2010.0108. Epub 2011 Feb 25. PMID 21352078
- [Background] Adeva MM, Souto G. Diet-induced metabolic acidosis. Clin Nutr. 2011 Aug;30(4):416-21. doi: 10.1016/j.clnu.2011.03.008. Epub 2011 Apr 9. PMID 21481501
- [Background] Samocha-Bonet D, Campbell LV, Mori TA, Croft KD, Greenfield JR, Turner N, Heilbronn LK. Overfeeding reduces insulin sensitivity and increases oxidative stress, without altering markers of mitochondrial content and function in humans. PLoS One. 2012;7(5):e36320. doi: 10.1371/journal.pone.0036320. Epub 2012 May 7. PMID 22586466
- [Background] Farwell WR, Taylor EN. Serum bicarbonate, anion gap and insulin resistance in the National Health and Nutrition Examination Survey. Diabet Med. 2008 Jul;25(7):798-804. doi: 10.1111/j.1464-5491.2008.02471.x. PMID 18644066
- [Background] Mandel EI, Curhan GC, Hu FB, Taylor EN. Plasma bicarbonate and risk of type 2 diabetes mellitus. CMAJ. 2012 Sep 18;184(13):E719-25. doi: 10.1503/cmaj.120438. Epub 2012 Jul 23. PMID 22825995
- [Background] Crawford SO, Hoogeveen RC, Brancati FL, Astor BC, Ballantyne CM, Schmidt MI, Young JH. Association of blood lactate with type 2 diabetes: the Atherosclerosis Risk in Communities Carotid MRI Study. Int J Epidemiol. 2010 Dec;39(6):1647-55. doi: 10.1093/ije/dyq126. Epub 2010 Aug 25. PMID 20797988
- [Background] Lovejoy J, Newby FD, Gebhart SS, DiGirolamo M. Insulin resistance in obesity is associated with elevated basal lactate levels and diminished lactate appearance following intravenous glucose and insulin. Metabolism. 1992 Jan;41(1):22-7. doi: 10.1016/0026-0495(92)90185-d. PMID 1538640
- [Background] Hayata H, Miyazaki H, Niisato N, Yokoyama N, Marunaka Y. Lowered extracellular pH is involved in the pathogenesis of skeletal muscle insulin resistance. Biochem Biophys Res Commun. 2014 Feb 28;445(1):170-4. doi: 10.1016/j.bbrc.2014.01.162. Epub 2014 Feb 3. PMID 24502946
- [Background] Akter S, Eguchi M, Kurotani K, Kochi T, Pham NM, Ito R, Kuwahara K, Tsuruoka H, Mizoue T, Kabe I, Nanri A. High dietary acid load is associated with increased prevalence of hypertension: the Furukawa Nutrition and Health Study. Nutrition. 2015 Feb;31(2):298-303. doi: 10.1016/j.nut.2014.07.007. Epub 2014 Jul 30. PMID 25592007
- [Background] Juraschek SP, Selvin E, Miller ER, Brancati FL, Young JH. Plasma lactate and diabetes risk in 8045 participants of the atherosclerosis risk in communities study. Ann Epidemiol. 2013 Dec;23(12):791-796.e4. doi: 10.1016/j.annepidem.2013.09.005. Epub 2013 Oct 5. PMID 24176820
- [Background] Heilbronn LK, Gan SK, Turner N, Campbell LV, Chisholm DJ. Markers of mitochondrial biogenesis and metabolism are lower in overweight and obese insulin-resistant subjects. J Clin Endocrinol Metab. 2007 Apr;92(4):1467-73. doi: 10.1210/jc.2006-2210. Epub 2007 Jan 23. PMID 17244782
- [Background] Maalouf NM, Cameron MA, Moe OW, Adams-Huet B, Sakhaee K. Low urine pH: a novel feature of the metabolic syndrome. Clin J Am Soc Nephrol. 2007 Sep;2(5):883-8. doi: 10.2215/CJN.00670207. Epub 2007 Aug 16. PMID 17702734